CLINICAL TRIAL: NCT01188811
Title: Lipoic Acid for Neuroprotection in Secondary Progressive MS
Brief Title: Lipoic Acid for Secondary Progressive Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7493-W
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Sclerosis, Chronic Progressive
Keywords: Multiple Sclerosis; Multiple sclerosis, chronic progressive; Neuroprotective agents; Magnetic resonance imaging; Optical coherence tomography; Gait; Thioctic acid; Alpha-lipoic acid
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: lipoic acid (Experimental): 28 subjects receive oral lipoic acid 1200mg daily
  Interventions: Drug: lipoic acid
- Arm 2: placebo (Placebo Comparator): 28 subjects receive placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lipoic acid — 1200 mg taken by mouth daily starting on day one of the study and ending on the last day of study participation.
  Other Names: alpha lipoic acid
  Arms: Arm 1: lipoic acid
Drug: Placebo — The placebo comparator will be taken by mouth daily starting on day one of the study and ending on the last day of study participation
  Arms: Arm 2: placebo

SUMMARY:
The purpose of the study is to determine if lipoic acid can protect the brain and slow disability in secondary progressive multiple sclerosis.

DETAILED DESCRIPTION:
There are no approved medications that are neuroprotective or able to slow disability accumulation in secondary progressive multiple sclerosis (SPMS). This two-year study will determine if daily oral intake of lipoic acid, a natural supplement, will prove superior to placebo in reducing injury to the brain and reducing disability progression in SPMS. Neuroprotection will be measured by the extent of brain volume loss seen on MRI, and disability will be measured by neurological status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SPMS
* Age 40-70 years
* Able to understand English and able to give informed consent

Exclusion Criteria:

* Unable to undergo MRI testing
* For ambulatory subjects only, a self-reported medical or neurological condition other than MS that is a cause of progressive or fluctuating problems that affect walking(e.g. worsening neuropathy, uncontrolled lower extremity arthritis, uncontrolled heart or lung disease)
* For ambulatory subjects only, fixed and/or stable conditions of less than 1 years duration that affect walking (e.g. joint replacement, lumbar stenosis, alcoholism, stroke, etc.)
* Pregnant or breast-feeding.
* Current major disease or disorder other than MS (such as cancer, kidney, heart or lung disease, post-traumatic stress disorder) that may interfere with study procedures
* Natalizumab, mitoxantrone, azathioprine taken in the last 12 months
* Other immunosuppressants or chemotherapies taken in the last 12 months
* Scheduled (every 3 months or more frequently) IV steroids used in the last 12 months
* IV or oral steroids taken in the past 60 days.
* Lipoic acid taken in the past 60 days.
* Subject has insulin-dependent diabetes or is not controlled on oral diabetes medications

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Spain, MD MSPH, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

REFERENCES:
- [Derived] Loy BD, Fling BW, Horak FB, Bourdette DN, Spain RI. Effects of lipoic acid on walking performance, gait, and balance in secondary progressive multiple sclerosis. Complement Ther Med. 2018 Dec;41:169-174. doi: 10.1016/j.ctim.2018.09.006. Epub 2018 Sep 22. PMID 30477834
- [Derived] Spain R, Powers K, Murchison C, Heriza E, Winges K, Yadav V, Cameron M, Kim E, Horak F, Simon J, Bourdette D. Lipoic acid in secondary progressive MS: A randomized controlled pilot trial. Neurol Neuroimmunol Neuroinflamm. 2017 Jun 28;4(5):e374. doi: 10.1212/NXI.0000000000000374. eCollection 2017 Sep. PMID 28680916

RESULTS

PARTICIPANT FLOW:
Groups:
- Lipoic Acid: 28 subjects receive oral lipoic acid 1200mg daily
  lipoic acid: 1200 mg taken by mouth daily starting on day one of the study and ending on the last day of study participation.
- Placebo: 28 subjects receive placebo daily
  Placebo: The placebo comparator will be taken by mouth daily starting on day one of the study and ending on the last day of study participation
Period: Overall Study
Arm/Group | Lipoic Acid | Placebo
Started | 28 | 26
Completed | 22 | 24
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lipoic Acid | Placebo | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 26 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (6.7) | 59.7 (6.1) | 58.7 (6.4)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Brain Atrophy by MRI
Time Frame: % change brain volume from baseline to year 2
Population: 22 subjects in the lipoic acid group and 24 in the placebo group completed the MRI outcome. Two outliers in the lipoic acid group were not included in analysis.
Measure: Mean (Standard Deviation); unit: whole brain percent volume change
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 20 | 24
whole brain percent volume change | -0.4 (0.7) | -1.3 (1.1)

2. Secondary Outcome: Disability Measures: Mobility
Time Frame: Change in Timed 25 Foot Walk from baseline to year 2
Population: Outliers were removed and intention-to-treat analysis was performed on data from 21 participants in the lipoic acid group and 17 in the placebo group.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 21 | 17
seconds | -1.0 (2.8) | 0.1 (2.0)

3. Secondary Outcome: Safety Measure: Adverse Events
Time Frame: adverse events recorded from baseline to year 2
Population: Intention-to-treat analysis was performed on 27 participants in the lipoic acid group and 24 in the placebo group.
Measure: Number; unit: occurences
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 27 | 24
occurences
  Total number adverse events | 81 | 69
  Total number serious adverse events | 9 | 6

ADVERSE EVENTS:
Arm/Group | Lipoic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 9/28 | 6/26
Other Adverse Events (participants affected / at risk) | 25/28 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipoic Acid (N=28) | Placebo (N=26)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CPK elevation (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipoic Acid (N=28) | Placebo (N=26)
Fall (Injury, poisoning and procedural complications) | 9 (11) | 13 (23)
Neoplasm: Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Spider Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Optic Neuritis (Eye disorders) | 1 (1) | 0 (0)
Peripapillary choroidal neovascularization (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gatroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI upset (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Edema of lower limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 3 (5) | 2 (2)
Gall bladder inflammation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Eye Infection (stye) (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 1 (1)
Oral ulcers (Infections and infestations) | 0 (0) | 1 (1)
Elevated Liver Enzymes (Investigations) | 1 (1) | 1 (1)
Otis externa (Infections and infestations) | 1 (1) | 0 (0)
Otis media (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 6 (8) | 8 (11)
Prostatitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 1 (1)
Vaginitis (Infections and infestations) | 0 (0) | 1 (1)
Varicella Zoster (Infections and infestations) | 1 (1) | 0 (0)
Viral Syndrome (Infections and infestations) | 1 (1) | 0 (0)
Abrasion (due to fall) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Left hand crush injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Left Knee Meniscus Tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Low WBC (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Right Knee) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysegusia (Nervous system disorders) | 1 (1) | 0 (0)
Face tingling/numbness (Nervous system disorders) | 0 (0) | 1 (1)
MS Relapse (Nervous system disorders) | 0 (0) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Kidney Stone with hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
nocturnal enuresis (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
rash (maculo-papular) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
surgical procedure- baclofen pump (Surgical and medical procedures) | 1 (1) | 0 (0)
Trigeminal neuralgia surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Benign nevi removed (Surgical and medical procedures) | 1 (1) | 0 (0)
Alkaline Phosphatase (Investigations) | 1 (1) | 0 (0)
Elevated creatinine (Investigations) | 1 (1) | 0 (0)
R. Eye Visual Sx (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No